CLINICAL TRIAL: NCT01626937
Title: Multicenter National Randomized Controlled Open Label Study Assessing Interest of Non Invasive Ventilation in out-of Hospital Setting During Acute Respiratory Failure in Chronic Obstructive Pulmonary Disease Patients. VeNIS BPCO
Acronym: VeNIS BPCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier d'Agen (Other)
Responsible Party: Principal Investigator, Pierre-Arnaud FORT, doctor, Centre Hospitalier d'Agen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A01382-39
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-01

CONDITIONS: Acute Respiratory Failure; Exacerbation of COPD; Non Invasive Positive Pressure Ventilation; Out of Hospital Setting
Keywords: Acute respiratory failure; Chronic obstructive pulmonary disease; Non invasive ventilation; Out of hospital
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

ARMS (2):
- Non invasive ventilation with conventional treatment (Experimental)
  Interventions: Other: Non invasive ventilation
- conventional medical treatment (Active Comparator)
  Interventions: Other: conventional medical treatment

INTERVENTIONS:
Other: Non invasive ventilation — After nebulisation of bronchodilatators and administration of corticosteroid therapy, non invasive positive pressure ventilation will be started out of hospital and continuously in COPD patient with acute respiratory distress and respiratory acidosis, using a facial mask, with initial level of inspiratory pressure at 8 mmHg then according to VTe and/or respiratory rate; expiratory pressure at 4 mmHg then according to persistance of inspiratory work, level of FiO2 for an objective of SpO2 between 88 and 92%. In case of failure, NIV will be stopped and endotracheal intubation realized if indicate.
  Arms: Non invasive ventilation with conventional treatment
Other: conventional medical treatment — Conventional medical treatment includes nebulization of bronchodilatators every 15-20 minutes until hospital and corticosteroid therapy. If indicate during out of hospital setting, endotracheale intubation will be realized. After admission in hospital, non invasive ventilation could be started.
  Arms: conventional medical treatment

SUMMARY:
Goal of the study: To show that prehospital NPPV use for COPD decompensation, as compared to only standard medical treatment, might enable a decrease in intubation rate.

Primary end point: the rate of endotracheal intubation in the first three hours after randomization.

Secondary en points: rate of endotracheal intubation after third hour, rate of prehospital and ICU mortality, ICU days, effects on clinical parameters (respiratory rate, SpO2, heart rate, arterial blood pressure, consciousness) and arterial blood gases (pH, PaCO2, PaO2), 30 days mortality, delays between first medical contact and in-hospital admission, relation between initial pH level and endotracheal intubation.

Inclusion criteria: Adult patients (>18 years), with GCS≥10, known or suspected COPD and presenting acute respiratory decompensation with respiratory acidosis.

Exclusion criteria: Cardiac or respiratory arrest, upper gastro intestinal tract haemorrhage, shock, serious ventricular arrhythmia, severe sepsis, multiple organ failure, serious cranial-facial trauma, upper airways obstruction, undrained pneumothorax, uncooperative-agitated patients refusing the technique, respiratory distress with bradypnoea < 12/min, pauses gasps repeated bradycardia, intractable vomiting, acute traumatic tetraplegia, persistant hemodynamic instability with PAS<90mmHg, ensuitable environment.

Randomization: Assignment to NPPV group or standard therapy group will be performed at the time of arrival of the SAMU team to the patient, by calling a physician located at the calldispatch center who will connect to the web site of the clinical research unit from Bordeaux university hospital.

Period of study: 25 months (24 months for patients inclusion and 1 month for follow-up).

Number of patients: 199 patients in each group i.e 398 patients (significance level of 5%, power of 80%; 50% expected decrease of intubation rate, i.e. from 20 to 10%).

Main investigator: Dr Pierre-Arnaud Fort, MD, Pôle Urgences-SAMU47-Réanimation, Centre Hospitalier Saint-Esprit - Agen.

Participating centers : 20 SAMU-SMUR corresponding to 19 departments in France.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years,
* Glasgow Coma Scale (GCS) ≥ 10,
* Written consent,
* Beneficiary social security regiment,
* Known or suspected COPD,
* Acute respiratory failure with FR > 25cycles/min,
* Setting concerned of the additional respiratory muscles and/or, paradoxical abdominal breathing,
* SpO2 < 90% with oxygen or decreasing rapidly under 90% with stop oxygen,
* PaCO2 > 45mmHg and pH < 7,35.

Exclusion Criteria:

* Cardiac or respiratory arrest,
* Upper gastro intestinal tract haemorrhage,
* Shock,
* Serious ventricular arrhythmia,
* Severe sepsis,
* Multiple organ failure,
* Serious cranial-facial trauma,
* Upper airways obstruction,
* Undrained pneumothorax,
* Uncooperative-agitated patients refusing the technique,
* Respiratory distress with bradypnoea < 12/min, pauses gasps repeated bradycardia,
* Intractable vomiting,
* Acute traumatic tetraplegia,
* Persistant hemodynamic instability with PAS<90mmHg,
* Ensuitable environment,
* Acute coronary syndrome,
* Serious acute asthma,
* Acute pulmonary edema,
* Acute respiratory insufficiency with lung before healthy,
* Gas of blood non available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
rate of endotracheal intubation in the first three hours after randomization | third hour after randomization

SECONDARY OUTCOMES:
rate of endotracheal intubation after third hour | after third hour during hospitalization